CLINICAL TRIAL: NCT06721923
Title: Continuous Versus Bolus Dietary Protein and Nutrition Status in the Pediatric Intensive Care Unit: Pilot Study
Brief Title: Continuous vs Bolus Protein (Protein Regimen Outcomes) in Critically Ill Children (Kids In Distress)
Acronym: PRO-KID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H23-00276
Record Dates: First submitted 2024-10-25; First posted 2024-12-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Critical Illness; Pediatric Intensive Care; Enteral Nutrition Therapy; Dietary Protein
Keywords: enteral nutrition; pediatric critical care; bolus protein delivery; continuous protein delivery; ultrasound; mid-upper arm circumference
MeSH Terms: conditions — Critical Illness | interventions — Dietary Proteins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous protein (Active Comparator): Continuous protein arm will have dietary protein supplement mixed into the enteral formula product to be provided around the clock without break.
  Interventions: Dietary Supplement: Dietary protein
- Bolus protein (Experimental): Bolus protein arm will provide protein powder mixed with water every 4h through syringe. This will be in addition to continuous enteral formula feeding which remains standard of care.
  Interventions: Dietary Supplement: Dietary protein

INTERVENTIONS:
Dietary Supplement: Dietary protein — Beneprotein powder, a whey-based supplement, will be used in both arms. Intervention dose will be 1g/kg of dietary protein (or 1.2g/kg of the powder), provided to both arms with different modes of delivery.

SUMMARY:
The goal of this intervention study is to evaluate the difference in nutrition status markers (weight and muscle mass) when giving dietary protein by continuous or bolus delivery in critically ill children ages 1-11y.

The main questions it aims to answer are:

Primary: Bolus protein delivery will lessen the decline in mid-upper arm circumference (MUAC) z-score by 0.5 standard deviation in critically ill children aged 1-11y after 1wk. Ultrasound will correlate to MUAC.

Secondary: Bolus protein delivery will provide more (grams per day) than when provided continuously, therefore it is more likely to meet the minimum estimated needs.

Participants will have daily nutrition intake data collected, and undergo body composition measures (weight, MUAC and ultrasound of the upper thigh muscle) at day of enrollment, and MUAC/Ultrasound on follow up days 3, 5, 7 and 14 after the intervention started.

DETAILED DESCRIPTION:
Daily screening and research advertisement posters will identify patients that may be eligible and interested in the study, this will be performed by the unit dietitian, research assistant or the physician/fellow (intensivist-trainee).The clinician dietitian who is the primary contact for the research study will not be involved outside the usual standard of care for patients in the pediatric intensive care unit (PICU). The following research steps will be completely by an established research team that is not directly involved in bedside care. Upon meeting inclusion criteria (age 1-11 years, expected length of stay >72h and enteral nutrition (EN) terminating in the stomach), informed consent will be presented verbally and in writing to the guardian present at bedside only if appropriate to approach the family during the early days (<48h) after admission. The research assistant or clinical nurse leader will review the project scope and any risks associated with participation with the family within 24-48 hours of admission if appropriate from a social and emotional viewpoint. For families that English is a second language, an interpreter will be used to provide information about the study and the consent details. Consent in escrow will be used for families admitted within traumatic circumstances where approaching research consent could cause undue stress to the guardians at bedside. The research team will have up to 14-days after admission to obtain written consent for the patients' data to be included in study analysis. Consent will be obtained or denied within 24 hours of presenting the study, or within 72 hours for deferred consent, after the formal conversation happens. All eligible patients will undergo non-invasive anthropometric assessment by trained professionals within 72 hours after admission to meet Assessment 0 criteria. Patients will be allocated into one of two intervention arms (continuous which is standard of care, or bolus) for supplemental protein delivery. We will allocate patients based on a blinded computer-generated draw utilizing block stratification for every 10 participants. Regular audits every 5 patients will allow evaluation of completed data so if one group appears to have more follow-up time points, the investigators will consult with the study team to determine whether temporary assignment into the underpowered group is required. Patients will be completely de-identified by research staff once data collection is complete to ensure no retrospective opinions or details are layered onto the result while data is being analyzed. Third-party statistician support will be sought out to further limit bias. Significant clinical changes, such as additional mechanical life support, will be noted to help enhance understanding and rationalize results when outcomes are discussed.

The intervention will begin after being prescribed the initial goal rate for continuous EN, this typically happens within the first 72-96 hours after admission. The clinical dietitian will be blinded to the treatment arm the patient has been allocated to. The online charting system will allow this blinding as the nursing view for accurate recording of patient care to be seen by the attending physicians is different from the allied health/dietitian view. All formulas are delivered continuously in our PICU, rarely would bolus feeds be started after a critical event. However, if this were the case the patient would not be eligible for study inclusion. Formula additives are prepared once a day by a centralized formula room. Given the restrictions around working hours, 24 hours to initiate intervention will be allowed to match typical operating procedure. Typically feeds/modules are ordered before 1200h, delivered around 1600h, and would be initiated shortly afterwards. The first day of the intervention will begin at 1900h to align with the units' feeding practices, nursing schedules, and online charting.

Protein dose will be held steady to ensure we are evaluating the mode of delivery and not the quantity of protein intake. We are aiming for a minimum intake of 2g/kg/day based off previous (2009) guidelines and our understanding of higher protein needs in a healthy population compared to current standards. The hypothesis that quality of protein delivery will improve uptake is why this pilot trial is not focusing on low versus high dosing. With previous research describing the theory of the "muscle full effect", we suspect patients may not need as high of a dose if protein is delivered more effectively. Based on a retrospective study in our unit, average protein intake is 0.8 - 1.6g/kg (SD 0.4) for patients 1-8 years old. Adding 1g/kg of supplemental protein will achieve 1.8-2.6g/kg/day which will allow us to meet the 2g/kg goal most of the time, while allowing us to focus on the feasibility and acceptance of the protein additive within the study context.

The continuous protein group will have 1g/kg of protein calculated and added into the formula which will continue to be delivered around the clock. Rate will be ordered as milliliters per hour with the expectation of running for 24 hours a day per standard care. The bolus protein group will be ordered 1g/kg protein to be divided and provided six times a day. The protein will remain separate from the formula, the latter will continue to be provided continuously per standard of care within the study unit. Protein will be provided every 4 hours to ensure ease of incorporating into standard nursing practice and individual medication schedule. Time of day the protein bolus is given, and amount will be recorded by the study team to ensure the daily target is achieved.

Study data will continue to be collected in our standardized forms if a patient is being fed exclusively through EN: the patient will be required to have continuous formula delivery and the protein intervention as set out at time of randomization. If either of these requirements is altered before 7 DPI, such as a change in continuous formula delivery to a different time schedule, if supplemental parenteral nutrition (PN) is initiation, or if the distal end of nutrition delivery is changed (from the stomach into the small bowel), the patient will no longer be eligible to have the protocolized protein intervention and the family will be notified as such. They may continue to receive supplemental protein; however, the schedule and amount will be based on the clinical judgement of the medical team/unit dietitian. Protein needs may become altered during admission, for example needing an increase in dose for evidence of delayed wound healing (open wounds or surgical sites), or if the consulting nephrologist wants to decrease protein load due to worsening kidney function: these adjustments will override the standard operating procedure for supplemental protein intervention. The energy prescription will be adjusted during the patients stay based on IC or energy equations and our understanding of the transition between acute to recovery phase nutrition requirements. This will not exclude patients from continuing with the study and data collection as long as any increase in energy needs, and total formula delivery, does not exceed the upper limit of protein dosing (4g/kg/day) which is called the renal solute load/limit. For the pilot trial we will note the length of intervention and follow up with the nutrition status assessments at the predetermined time points. The duration of intervention will be included in statistical analysis. Transition to a more appropriate EN regime will not be prevented due to study participation.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to PICU over 1 year of age and younger than 11 years of life
* Expected to remain in the pediatric intensive care unit for longer than 72 hours
* Receiving standard pediatric formula via NGT/OGT/GT

Exclusion Criteria:

* Neuromuscular condition such as muscular dystrophy
* Admitted with home prescription for high dose steroids, receives growth hormone or insulin
* Enteral nutrition is contraindicated or if nutrition requirements are partially/fully met by parenteral nutrition
* Formula delivered into the small bowel (duodenum/jejunum, NJT/GJ)
* Those who require a highly specialized diet (E.g., large burns or metabolic diseases)
* Patients with a cow's milk protein allergy cannot safely receive a whey-based protein supplement

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Mid-upper arm circumference | admission, 7 and 14 days
  Mid-upper arm circumference (MUAC) will be the primary outcome measure with a standard deviation change in z-score of 0.5 being considered significant. The measure (in centimeters) will be assessed against the WHO validated growth standard (for sex and age) and reported as z-score to standardized the measures against the population as a whole.

SECONDARY OUTCOMES:
Ultrasound of the Rectus Femoris Quadricep | admission, 7 and 14 days
  Ultrasound of the upper thigh (quadricep) muscle (rectus femoris) will be used (in centimeters) to compare with MUAC (in centimeters) and protein delivery (grams per day and percentage of minimum intake). This will be an exploratory measurement to detect the percentage change over time between ultrasound and MUAC. It will then be explored whether both protein groups (continuous vs bolus) have a similar change in percentage over time.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — University of British Columbia, Department of Pediatrics
Locations (1):
- BC Childrens Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
At this time we are performing pilot work and have indicated to ethics this was not the intention of this work.

REFERENCES:
- [Background] El-Kadi SW, Boutry C, Suryawan A, Gazzaneo MC, Orellana RA, Srivastava N, Nguyen HV, Kimball SR, Fiorotto ML, Davis TA. Intermittent bolus feeding promotes greater lean growth than continuous feeding in a neonatal piglet model. Am J Clin Nutr. 2018 Oct 1;108(4):830-841. doi: 10.1093/ajcn/nqy133. PMID 30239549
- [Background] Davis TA, Fiorotto ML, Suryawan A. Bolus vs. continuous feeding to optimize anabolism in neonates. Curr Opin Clin Nutr Metab Care. 2015 Jan;18(1):102-8. doi: 10.1097/MCO.0000000000000128. PMID 25474017
- [Background] Rudar M, Naberhuis JK, Suryawan A, Nguyen HV, Stoll B, Style CC, Verla MA, Olutoye OO, Burrin DG, Fiorotto ML, Davis TA. Intermittent bolus feeding does not enhance protein synthesis, myonuclear accretion, or lean growth more than continuous feeding in a premature piglet model. Am J Physiol Endocrinol Metab. 2021 Dec 1;321(6):E737-E752. doi: 10.1152/ajpendo.00236.2021. Epub 2021 Nov 1. PMID 34719946
- [Background] Ong C, Lee JH, Senna S, Chia AZH, Wong JJM, Fortier MV, Leow MKS, Puthucheary ZA. Body Composition and Acquired Functional Impairment in Survivors of Pediatric Critical Illness. Crit Care Med. 2019 Jun;47(6):e445-e453. doi: 10.1097/CCM.0000000000003720. PMID 30958426
- [Background] Ong C, Lee JH, Wong JJM, Leow MKS, Puthucheary ZA. Skeletal Muscle Changes, Function, and Health-Related Quality of Life in Survivors of Pediatric Critical Illness. Crit Care Med. 2021 Sep 1;49(9):1547-1557. doi: 10.1097/CCM.0000000000004970. PMID 33861558
- [Background] Valverde Montoro D, Rosa Camacho V, Artacho Gonzalez L, Camacho Alonso JM. Thigh ultrasound monitoring identifies muscle atrophy in mechanically ventilated pediatric patients. Eur J Pediatr. 2023 Dec;182(12):5543-5551. doi: 10.1007/s00431-023-05233-4. Epub 2023 Oct 2. PMID 37782351
- [Background] Hulst JM, Huysentruyt K, Gerasimidis K, Shamir R, Koletzko B, Chourdakis M, Fewtrell M, Joosten KF; Special Interest Group Clinical Malnutrition of ESPGHAN. A Practical Approach to Identifying Pediatric Disease-Associated Undernutrition: A Position Statement from the ESPGHAN Special Interest Group on Clinical Malnutrition. J Pediatr Gastroenterol Nutr. 2022 May 1;74(5):693-705. doi: 10.1097/MPG.0000000000003437. Epub 2022 Mar 3. PMID 35258497
- [Background] Becker P, Carney LN, Corkins MR, Monczka J, Smith E, Smith SE, Spear BA, White JV; Academy of Nutrition and Dietetics; American Society for Parenteral and Enteral Nutrition. Consensus statement of the Academy of Nutrition and Dietetics/American Society for Parenteral and Enteral Nutrition: indicators recommended for the identification and documentation of pediatric malnutrition (undernutrition). Nutr Clin Pract. 2015 Feb;30(1):147-61. doi: 10.1177/0884533614557642. Epub 2014 Nov 24. PMID 25422273